CLINICAL TRIAL: NCT02985463
Title: Left Atrial Appendage Occlusion and Biomarker Evaluation
Acronym: LABEL
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Universitätsmedizin Mannheim (Other)
Responsible Party: Principal Investigator, Michael Behnes, Dr. med, Universitätsmedizin Mannheim
Other Study IDs: 2014-402M-MA-§ 23b MPG
Record Dates: First submitted 2016-12-03; First posted 2016-12-07 (Estimated); Last update posted 2020-08-27 (Actual); Status verified 2020-08

CONDITIONS: Stroke; Atrial Fibrillation; Bleeding
MeSH Terms: conditions — Stroke; Atrial Fibrillation; Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Two peripheral blood withdraws in EDTA, citrate, ammonium heparin, serum tubes 24 hours before and at mid-term follow up at 6 months after successful LAA occlusion device implantation.
Oversight: Data Monitoring Committee: No

SUMMARY:
"Left Atrial Appendage Occlusion and Biomarker Evaluation" (LABEL) is a single-center, prospective and observational study evaluating changes of the expression of biomarkers in eligible patients before and after percutaneous implantation of a left atrial appendage (LAA) occlusion device at mid-term follow-up.

DETAILED DESCRIPTION:
This study will evaluate the changes of different types of biomarkers before and after successful percutaneous implantation of an LAA occlusion device.

Biomarker evaluation will focus on blood derived biomarkers including neurohormones, proteins, cytokines, microRNAs and metabolomics.

ELIGIBILITY:
Inclusion Criteria:

* non valvular atrial fibrillation, that makes anticoagulation to prevent embolic stroke from the LAA
* contraindication for the therapy with oral anticoagulants:
* refusal to take oral anticoagulation
* HasBled-score more than 3
* prior bleedings under oral anticoagulation

Exclusion Criteria:

* under 18 years
* severely reduced left atrial function
* mechanical heart valve
* pulmonary embolism
* deep vein thrombosis
* myocardial infarction within the last 3 months
* electrical cardioversion within 30 days after potential occluder implantation
* atrial septum defect or interventional/surgical occlusion of ASD
* status after heart transplant
* symptomatic carotid artery stenosis
* transient ischemic attack (TIA) or stroke within last 30 days
* intracerebral bleeding within the last 2 months
* acute infection
* existing or planned pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients suffering from non valvular atrial fibrillation with a contraindication for oral anticoagulation (i.e. bleeding) being eligible of percutaneous implantation of LAA occlusion devices.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2014-06 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Biomarker levels before successful LAA occlusion device implantation | 24 hours before intervention

SECONDARY OUTCOMES:
Biomarker levels after successful LAA occlusion device implantation | mid-term follow up at 6 months
Changes of biomarker expression before and after device implantation over mid-term follow-up, depending of complete, incomplete occlusion, imaging data (transesophageal echocardiography, computed tomography) | mid-term follow up at 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Ibrahim Akin, Prof., Study Director — University Medical Center Mannheim
Locations (1):
- University Medical Centre Mannheim, Mannheim, Baden-Wurttemberg, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Behnes M, Akin I, Sartorius B, Fastner C, El-Battrawy I, Borggrefe M, Haubenreisser H, Meyer M, Schoenberg SO, Henzler T. --LAA Occluder View for post-implantation Evaluation (LOVE)--standardized imaging proposal evaluating implanted left atrial appendage occlusion devices by cardiac computed tomography. BMC Med Imaging. 2016 Mar 24;16:25. doi: 10.1186/s12880-016-0127-y. PMID 27009279
- [Result] Fastner C, Behnes M, Sartorius B, Yildiz M, Mashayekhi K, El-Battrawy I, Lehmann R, Baumann S, Becher T, Borggrefe M, Akin I. Left atrial appendage morphology, echocardiographic characterization, procedural data and in-hospital outcome of patients receiving left atrial appendage occlusion device implantation: a prospective observational study. BMC Cardiovasc Disord. 2016 Jan 28;16:25. doi: 10.1186/s12872-016-0200-z. PMID 26822890
- [Derived] Rusnak J, Behnes M, Saleh A, Fastner C, Sattler K, Barth C, Wenke A, Sartorius B, Mashayekhi K, Hoffmann U, Yuecel G, Lang S, Borggrefe M, Akin I. Interventional left atrial appendage closure may affect metabolism of essential amino acids and bioenergetic efficacy. Int J Cardiol. 2018 Oct 1;268:125-131. doi: 10.1016/j.ijcard.2018.05.031. Epub 2018 Jun 1. PMID 29861102
- [Derived] Fastner C, Behnes M, Sartorius B, Wenke A, Lang S, Yucel G, Sattler K, Rusnak J, Saleh A, Barth C, Mashayekhi K, Hoffmann U, Borggrefe M, Akin I. Interventional Left Atrial Appendage Closure Affects the Metabolism of Acylcarnitines. Int J Mol Sci. 2018 Feb 7;19(2):500. doi: 10.3390/ijms19020500. PMID 29414920